CLINICAL TRIAL: NCT01768104
Title: Endoscopic Submucosal Tunnel Dissection Versus Video-assisted Thoracoscopic Surgery for Upper Gastrointestinal Submucosal Tumors: a Prospective Randomized Controlled Trial
Brief Title: ESTD vs. VATS for Upper Gastrointestinal Submucosal Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFEK-201211-K1; 201120 (Other Grant/Funding Number: New business and New Technology Project of Nanfang Hospital)
Record Dates: First submitted 2013-01-05; First posted 2013-01-15 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2011-12

CONDITIONS: Upper Gastrointestinal Submucosal Tumors (SMTs); Gastrointestinal Stromal Tumors (GISTs); Leiomyoma
Keywords: upper gastrointestinal submucosal tumors; SMTs; Gastrointestinal stromal tumors; GISTs; Leiomyoma; Endoscopic submucosal tunnel dissection; ESTD; Submucosal tunneling endoscopic resection; STER; Submucosal endoscopic tumor resection; SET
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Leiomyoma | interventions — Endoscopic Mucosal Resection; Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ESTD (Experimental): Endoscopic submucosal tunnel dissection (ESTD) for patients with upper gastrointestinal submucosal tumors (SMTs)
  Interventions: Procedure: ESTD
- VATS (Active Comparator): Video-assisted thoracoscopic surgery (VATS) for patients with upper gastrointestinal submucosal tumors (SMTs)
  Interventions: Procedure: VATS

INTERVENTIONS:
Procedure: ESTD — 1. A 2-cm longitudinal mucosal incision was made, approximately 5cm proximal to the submucosal tumor (SMTs).
  2. Submucosal dissection was done, creating a submucosal tunnel until the tumor was visible.
  3. Dissection was done along the margin of the tumor.
  4. After the tumor had been removed, the potential bleeding area in the tunnel was coagulated.
  5. Endoclips were used to close the entry of the submucosal tunnel.
  (Gong W et al. ESTD for upper gastrointestinal submucosal tumors… Endoscopy 2012; 44: 231-235)
  Other Names: Endoscopic submucosal tunnel dissection (ESTD); Submucosal tunneling endoscopic resection (STER); Submucosal endoscopic tumor resection (SET)
  Arms: ESTD
Procedure: VATS — 1. General anesthesia with double lumen intubation.
  2. Three to four cameras or working ports are placed over the chest wall.
  3. After the lesion is visualized by thoracoscopy, the mediastinal pleura over the tumor is incised longitudinally by an endoscopic hook electrocauterizer.
  4. The mass is exposed after the overlying muscle is split longitudinally.
  5. The retracting suture is placed over the mass and then meticulously dissect the plane between the mass and the submucosal layer. The integrity of the mucosa must be checked.
  6. The muscle layer is re-approximated and a chest tube is place through one of the ports.
  (Luh et al. World Journal of Surgical Oncology 2012, 10:52)
  Other Names: Video-assisted thoracoscopic surgery; Video-thoracoscopic enucleation
  Arms: VATS

SUMMARY:
The purpose of this study is to determine the efficacy and safety of endoscopic submucosal tunnel dissection (ESTD) compared with video-assisted thoracoscopic surgery (VATS) in the treatment of upper gastrointestinal submucosal tumors.

DETAILED DESCRIPTION:
Most upper gastrointestinal submucosal tumors (SMTs), especially the gastrointestinal stromal tumors (GISTs) and leiomyoma, are regarded as benign if they are less than 3cm in size. Thus, it has been suggested that patients should receive periodic endoscopic follow-up in case of gradual changes in size; however this can be stressful and troublesome for patients. Nevertheless, some of these tumors do have a malignant potential, and management by periodic endoscopic surveillance may lead to delayed diagnosis of malignancy. Therefore, it is necessary to remove the SMTs.

To date, several approaches have been used for the treatment of upper gastrointestinal SMTs, including open, thoracoscopic and laparoscopic surgery, and endoscopic approaches such as band ligation, endoscopic submucosal dissection (ESD), and endoscopic full-thickness resection (EFR). However, the surgical approaches are invasive with a longer hospital stay and greater cost, while the endoscopic approaches were limited by technical difficulty, incomplete resections and risk of perforation.

Recently, the technique of peroral endoscopic myotomy (POEM) for esophageal achalasia was introduced, a procedure in which a submucosal tunnel is created to expose and dissect the circular muscle of the esophagus. Inspired by the POEM approach, we have successfully used a similar method, endoscopic submucosal tunnel dissection (ESTD), to resect SMTs in upper gastrointestinal.

However, the long-term efficacy and safety of ESTD were not determined, and there was no prospective study compared the ESTD with other conventional approaches. Therefore, we plan to conduct this prospective randomized controlled trial, aim to determine the efficacy and safety of ESTD, compared with the pneumatic dilation, in the treatment of upper gastrointestinal SMTs originating from the muscularis propria layer .

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 75 years of age
* Patient with upper gastrointestinal submucosal tumor
* Signed informed consent

Exclusion Criteria:

* Severe cardio-pulmonary disease or other serious disease leading to unacceptable surgical risk
* Endoscopic ultrasound (EUS) or CT signs of metastasis
* Mega-oesophagus (greater than 7 cm) or Oesophageal diverticula in the distal oesophagus
* Previous oesophageal or gastric surgery
* Pregnancy or lactation women, or ready to pregnant women
* Not capable of filling out questionnaires

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
En bloc resection | During the operation
  The En bloc resection was defined as a one-piece resection of the entire lesion without fragmentation

SECONDARY OUTCOMES:
Curative resection | From date of randomization until the date of pathological diagnosis, an expected average of 7 days
  The curative resection was defined as the resected specimen with vertical and lateral margins free of neoplasia in pathological diagnosis.
Procedure related complication | From date of operation until the occurrence of the procedure related complication, which most occur within 7 days after operation, assessed up to 2 years
  Perforation, Delayed bleeding, Pneumothorax, Subcutaneous emphysema, Anastomotic leak, etc.
Short-term morbidity | From date of randomization until the date of death from any cause, assessed up to 3 months
  Any cause death
Local recurrence | From date of randomization until the follow-up ended, assessed up to 2 years
  Local recurrence was defined as endoscopic or histological diagnosis of cancer at the resected site in follow-up
Quality of life | From date of randomization until the follow-up ended, assessed up to 2 years
  Patients will complete the quality-of-life questionnaires (the Medical Outcomes Study 36-Item Short-Form Health Survey, SF-36) for assessing quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Wei Gong, M.D., Principal Investigator — Department of Gastroenterology, Nanfang Hospital of Southern Medical University
Locations (1):
- Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Gong W, Xiong Y, Zhi F, Liu S, Wang A, Jiang B. Preliminary experience of endoscopic submucosal tunnel dissection for upper gastrointestinal submucosal tumors. Endoscopy. 2012 Mar;44(3):231-5. doi: 10.1055/s-0031-1291720. Epub 2012 Feb 21. PMID 22354823
- [Background] Zhao Y, Cai K, Liu D, Wu H, Xiong G, Wang H, Huang Z, Cai R, Wu X. [Video-assisted thoracoscopic removal of esophageal leiomyomas with intraoperative tumor location by endoscopy]. Nan Fang Yi Ke Da Xue Xue Bao. 2012 Apr;32(4):586-8. Chinese. PMID 22543150
- See also: Homepage of Nanfang Hospital of Southern Medical University — http://www.nfyy.com/
- See also: Homepage of Department of Gastroenterology, Nanfang Hospital of Southern Medical University — http://www.xhbnet.com/